CLINICAL TRIAL: NCT00968188
Title: A Randomized Control Trial of an Internet-based HIV/STI Prevention for Young MSM Receiving HIV Testing.
Brief Title: Internet-based HIV/STI Prevention for Young MSM Receiving HIV Testing
Acronym: KIU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Brian Mustanski, PhD / Assistant Professor and Director, IMPACT Program, University of Illinois at Chicago, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2007-0182; 1R34MH079714-01A1 (NIH)
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: HIV; HIV Infections
Keywords: HIV Risk; Internet Intervention; Homosexuality, Male; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Homosexuality, Male

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active intervention (Experimental): Highly interactive, motivational, culturally tailored, online HIV prevention.
  Interventions: Behavioral: Keep It Up!
- Information only (Active Comparator): Medically fact based online intervention.
  Interventions: Behavioral: Information only

INTERVENTIONS:
Behavioral: Keep It Up! — Online HIV Intervention Prevention Website tailored to Young Men that Have Sex with Men. Website is tailored to be more engaging, includes videos and games.
  Arms: Active intervention
Behavioral: Information only — Medically fact based HIV information delivered online.
  Arms: Information only

SUMMARY:
The purpose of this study is to develop an empirically validated, scientifically-based HIV and STI prevention program that can be delivered online to young men who have sex with men (YMSM) who were recently tested for HIV.

DETAILED DESCRIPTION:
Presently, there are a limited number of proven HIV interventions culturally tailored to young men who have sex with men (YMSM). This is alarming because Men who have sex with men comprise 68% of HIV/AIDS diagnoses in men, despite representing a much smaller proportion of the population. In addition, MSM are reporting more sexual risk behavior than in previous years and there is significant concern that HIV infection rates may once again be on the rise after more than a decade of remaining relatively stable.

The Internet is a viable intervention avenue because of it's high percentage of accessibility and usage, especially among young adults. Moreover, it might hold a strong appeal for YMSM, since its anonymity confers a sense of perceived safety against stigma surrounding HIV prevention information.

The purpose of this study is to compare two different versions of an online HIV/STI intervention for YMSM. This study is part of an overall program of research designed to understand and prevent HIV infection among high-risk youth. Participation in this study will help us to determine the usefulness of an tailored and interactive HIV Internet-assisted intervention.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 24 years of age
* Self-identify as a biological male
* Understand and read English
* Have tested HIV negative at an approved clinic within 6 weeks
* Report at least one (male) sex partners in the past three months, and unprotected anal sex with at least one male sex partner in the past three months.

Exclusion Criteria:

* Have been diagnosed with HIV within the past three months
* Participation in another HIV prevention program
* No access to the Internet or an email address

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Sexual Risk Behavior | 3 months

SECONDARY OUTCOMES:
HIV knowledge, Decisional Balance, condom errors, safer sex self-efficacy, intentions | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian S Mustanski, PhD, Principal Investigator — Northwestern University
Locations (1):
- Howard Brown Health Center, Chicago, Illinois, United States